CLINICAL TRIAL: NCT03986619
Title: Evaluation of Methods for Measuring Food Reward and Food-related Behavior in Healthy Individuals - a Substudy of the PRESET Study
Brief Title: Evaluation of Methods for Measuring Food Reward and Food-related Behavior in Healthy Individuals
Acronym: PRESET
Status: Completed | Type: Observational
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Copenhagen (Other); University of Leeds (Other); Aalborg University Hospital (Other); IMotions A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: H-18026293_substudy
Record Dates: First submitted 2019-06-06; First posted 2019-06-14 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Healthy Participants
Keywords: Food preferences; Food reward
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most of the decisions and actions affecting energy balance are driven by implicit and explicit motivational processes. In modern obesogenic environment where highly palatable and energy-dense foods are easily available, it is of great interest to increase the understanding of both implicit and explicit processes of food-related behavior.

The aim of the present study is to examine whether biometric signatures in response to visual food stimuli during the already validated Leeds Food Preference Questionnaire (LFPQ) correlate with liking, wanting, food choice, or subsequent ad libitum food intake of those foods as assessed by the LFPQ and an ad libitum buffet meal.

DETAILED DESCRIPTION:
Human behaviour including food reward plays a pivotal role in appetite regulation and the type and amount of food eaten. Food reward is a driver of eating behaviour and is defined as the momentary value of a food to the individual at the time of ingestion. Food reward contains the components of liking and wanting that can exist both with (explicit) and without (implicit) conscious awareness. Most of the daily decisions and actions affecting energy balance are driven by the non-conscious mind. Non-conscious processes are characterised by being unintentional and without awareness of the effects of triggering stimuli, e.g. food items. Contrary, conscious processes are typically assessed through participants' self-reports but limited by accuracy and desire to provide socially desirable answers. In a world of plenty where foods are always easily available with an overtly representation of highly palatable and energy-dense foods it is of great interest to understand the role of the non-conscious mind as a driver of food choice and intake. Intake of highly palatable and energy-dense foods is related to excess energy intake, high body mass index and weight gain. A possible explanation for this is that these foods are overall more rewarding and as a result of this, palatable.

A few previous studies have applied the use of innovative biometric measures, i.e. eye tracking, galvanic skin response, and facial expression to examine behavioural aspects of food intake that are without conscious awareness. However, there is a lack of studies examining how biometric responses to different food groups varying in energy density and palatability correlate with outcomes related to components of food reward and food intake. Therefore, in the present explorative study the above-mentioned biometric measurements will be combined with an existing validated method, the Leeds Food Preference Questionnaire (LFPQ), developed to examine both non-conscious and conscious components of food reward. The LFPQ assess four factors related to food reward within four combined food categories: food choice, implicit and explicit wanting, and explicit liking for high-fat sweet foods, low-fat sweet foods, high-fat savoury foods, and low-fat savoury foods. Biometric measurements of eye tracking can provide measures of attention, measurements of galvanic skin response can provide measures of arousal, and facial expressions analyses can provide information on emotional responses in response to selected stimuli, which in this study constitute pictures of food items. Furthermore, the study will include a taste task including an ad libitum intake of test foods in order to examine responses to actual food intake and to compare these responses to biometric responses to visual food stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Age: from ≥30 to ≤70 years of age
* BMI: from 18.5 to 24.9 kg/m2

Exclusion Criteria:

* Unable to understand the informed consent and the study procedures;
* Allergic to the food items included in the taste test
* Self-reported history of an eating disorder in the past three years
* Self-reported weight change (>5 kg) within three months prior to inclusion

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal-weight individuals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Gaze duration bias (ratio) | 0 minutes (fasting)
  A measure of attention measured using eye tracking in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire.
  Gaze duration bias is calculated as the average gaze duration (ms) to a specific food image relative to the average gaze duration to all images.
  A bias score ˃0.5 indicates maintained attention towards a food image, a bias score equal to 0.5 indicates no bias, and a bias score <0.5 indicates maintained attention towards the other food images.

SECONDARY OUTCOMES:
Attention | 0 minutes (fasting)
  Measured using eye tracking in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire.
  Includes the following parameters: Gaze: Time spent (ms and %) and revisits (n); and fixations: Time to first fixation (ms), time spent (ms and %), fixation count (n), first fixation duration (ms), average fixation duration (ms). Distance to screen (mm), and gaze direction bias (ratio) which is calculated as the number of trials in which the first fixation was directed to a food image as a proportion to all trials. A bias score ˃0.5 indicates attention towards one food image, a bias score equal to 0.5 indicates no bias, and a bias score <0.5 indicates attention towards the other food images.
Arousal | 0 minutes (fasting)
  Measured as galvanic skin response (changes in conductivity of the skin) in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire.
  Includes the following parameters: Presence of a peak (yes/no), peak count (n), peaks/min, peak (ms), peak amplitude (μS), peak onset (ms), peak offset (ms), duration (ms), tonic signal (μS).
  The presence of a peak, the magnitude of the peak as well as the duration of the peak are measures of arousal (includes all the parameters listed above). The greater the response the higher the arousal.
Emotions | 0 minutes (fasting)
  Emotions including anger, sadness, disgust, joy, surprise, fear, contempt as well as facial expression metrics (actions units) are determined by facial expression analysis using computer-vision algorithms (AFFDEX) in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire.
  Results represent the probability the emotions and facial expression metrics were expressed (range: 0-100; 0=it was not expressed, 100=it was expressed, 50=50% likelihood that it was expressed).
Food choice | 0 minutes (fasting)
  Food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Food choice is determined based on frequency of selection made within each food category. The scores range from 0-48 i.e. 0 = foods within a specific food category have not been selected at all to 48 = foods within a specific food category have been selected 48 times.
Reaction time (ms) | 0 minutes (fasting)
  Reaction time during forced food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire.
Implicit wanting | 0 minutes (fasting)
  Implicit wanting of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Implicit wanting is assessed based on food choice and response time for selected and non-selected food items as well as mean response time (a frequency-weighted algorithm).
  In this frequency-weighted algorithm a positive score indicates a more rapid preference for a food type over another food type and a negative score indicates the opposite. A score of zero indicates that food types are equally preferred. The frequency weighted algorithm is used so the implicit wanting score is influenced by both selection (positively contributing to the score) and non-selection (negatively contributing to the score) of food type. Scores for implicit wanting typically range from -100-100 (due to reaction time there is no fixed min-max value)
Explicit liking | 0 minutes (fasting)
  Explicit liking of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Explicit liking is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how pleasant would it be to taste this food right now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Explicit wanting | 0 minutes (fasting)
  Explicit wanting of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire. Explicit wanting is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how much do you want some of this food now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Subjective appetite | 0 minutes (fasting)
  Rated using visual analogue scales and includes sensations of: Hunger, fullness, satiety, prospective food consumption, wellbeing, nausea, thirst, desire to eat meat, salty, and sweet. The scale range is 0-100 and each end represent the extremes e.g. hunger rating: "I am not hungry at all" to "I have never been this hungry before".
Body weight (kg) | 0 minutes (fasting)
  Body weight is measured on a digital scale
Body mass index (kg/m^2) | 0 minutes (fasting)
  Calculated from body weight (kg) and height (m)
Fat mass (kg) | 0 minutes (fasting)
  Measured by Dual-energy X-ray Absorptiometry
Fat percentage (%) | 0 minutes (fasting)
  Measured by Dual-energy X-ray Absorptiometry
Fat free mass (kg) | 0 minutes (fasting)
  Measured by Dual-energy X-ray Absorptiometry
Waist circumference (cm) | 0 minutes (fasting)
  Measured using tape measure
Hip circumference (cm) | 0 minutes (fasting)
  Measured using tape measure
Systolic blood pressure (mmHg) | 0 minutes (fasting)
  Measured under resting and fasting conditions
Diastolic blood pressure (mmHg) | 0 minutes (fasting)
  Measured under resting and fasting conditions
Heart rate (bpm) | 0 minutes (fasting)
  Measured under resting and fasting conditions
HbA1c (mmol/mol and %) | 0 minutes (fasting)
  Hemoglobin A1c
Sleep quality | 0 minutes (fasting)
  Assessed using the Pittsburgh Sleep Quality Index. The questionnaire covers sleep quality and sleep disturbances over the preceding month and includes 19 individual items that generate seven scores weighted on a 0-3 scale. The sum of the component scores yields a total score of 0-21, and the higher the score, the poorer the sleep quality. The questionnaire also covers bedtime (hh:mm), sleep onset latency (minutes/night), wake-up (hh:mm); sleep duration (hours and minutes per night).
Sleepiness | 0 minutes (fasting)
  Assessed using the Epworth Sleepiness Scale. The questionnaire describes eight different situations of everyday life, and participants are asked to rate how likely they would doze off or fall asleep in each situation on a 0-3 scale. The sum of the scores yields a total score of 0-24, with higher scores indicative of greater daytime sleepiness.
Self-reported health | 0 minutes (fasting)
  Assessed using the Short Form Health Survey (SF-36). The questionnaire covers self-reported health status and the response format is a Likert-type scale e.g. question regarding overall health from 1=excellent to 5=poor and binary scales (yes/no) e.g. "difficulties performing daily tasks".
Physical activity | Minimum 6 hours after test day
  Assessed using the Recent Physical Activity Questionnaire. The questionnaire covers physical activity during work and in transport and leisure-time domains. The response format is a Likert-type scale e.g. 1=never and 5=always and participants are also asked about distance to work and typical mode of transportation. The time spent (minutes/day) on different modes of transportation or work-related or leisure-time physical activities and exercise as well as intensity (sedentary, light, moderate, vigorous) of the activities can be calculated.
Chronotype | 0 minutes (fasting)
  Assessed using the Munich Chronotype Questionnaire. The primary outcome is sleep midpoint (hh:mm) calculated based on participants' registration of habitual bedtime (hh:mm), sleep onset (hh:mm), sleep onset latency (minutes), wake-up (hh:mm), time from wake-up to out of bed (minutes). The questionnaire also covers use of sleep medicine and intake of alcohol and coffee/tea (units/day, units/ week, units/months), type of transportation to work (car/bus/train, walking/bicycling or work from home) and duration of transportation (minutes/day).
Night eating | Minimum 6 hours after test day
  Assessed using the Night Eating Questionnaire. The questionnaire covers hunger and craving for foods at different times during the day and night. The response format is a Likert-type scale ranging from e.g. 0=not at all to 4=very much.
Eating behavior | Minimum 6 hours after test day
  Assessed using the Dutch Eating Behavior Questionnaire. The questionnaire consists of 33 questions and assess restrained (10 items), emotional (13 item), and external (10 items) eating behavior. The response format is a Likert-type scale ranging from 1=never to 5= very often. The greater the total score within each category the greater degree of e.g. dietary restraint.
Control over eating | Minimum 6 hours after test day
  Assessed using the Control Over Eating Questionnaire. Control of eating and the degree of food cravings are assessed using the 21-item questionnaire which includes questions related to food cravings, control of eating, appetite and overall mood. Based on the previous 7 days, participants are asked to rate 20 questions on a 100 mm visual analogue scale (VAS). One question is open-ended. The VAS range is 0-100 and each end represent the extremes e.g. "how difficult is it to control eating": "Not difficult at all" to "It has never been more difficult".
Socioeconomic status | 0 minutes (fasting)
  Assessed using a questionnaire assessing self-reported educational level (categorical), main occupation (categorical), civil status (categorical), ethnicity (categorical), living arrangement (categorical), children (n), personal income (DKK), household income (DKK), sex (male/female), and age (years).
Total energy intake (kcal or kJ) | 60 minutes after basal assessments
  Total energy intake during an ad libitum buffet meal provided after all basal assessments
Energy intake from specific food categories (kcal or kJ) | 60 minutes after basal assessments
  Energy intake from different food categories (high fat-savoury, high fat-sweet, low fat-savoury, low fat-sweet) during an ad libitum buffet meal provided after all basal assessments
Explicit liking | 60 minutes after basal assessments
  Explicit liking of 8 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined during an ad libitum buffet meal provided after all basal assessments. Explicit liking is rated using visual analogue scales and the range is 0-100. Each end represents the extremes. Question: "how pleasant is the taste of the food right now?" Answer: "not pleasant at all" (rated 0 on the 0-100 scale) to "very pleasant" (rated 100 on the 0-100 scale).
Explicit wanting | 60 minutes after basal assessments
  Explicit wanting of 8 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined during ad libitum buffet meal provided after all basal assessments. Explicit wanting is rated using visual analogue scales and the range is 0-100. Each end represents the extremes. Question: "How much more do you think you can eat of the food right now?" Answer: "nothing at all" (rated 0 on the 0-100 scale) to "very much" (rated 100 on the 0-100 scale).

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Færch, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Pedersen H, Diaz LJ, Clemmensen KKB, Jensen MM, Jorgensen ME, Finlayson G, Quist JS, Vistisen D, Faerch K. Predicting Food Intake from Food Reward and Biometric Responses to Food Cues in Adults with Normal Weight Using Machine Learning. J Nutr. 2022 Jun 9;152(6):1574-1581. doi: 10.1093/jn/nxac053. PMID 35325189